CLINICAL TRIAL: NCT06055465
Title: Neoadjuvant Sacituzumab Govitecan Plus Pembrolizumab in Resectable Non-Small Cell Lung Cancer: an Open-label, Multicenter, Single Arm Phase 2 Study
Brief Title: Neoadjuvant Sacituzumab Govitecan Plus Pembrolizumab in Resectable Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Molly SC Li, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUN109
Record Dates: First submitted 2023-08-24; First posted 2023-09-26 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — sacituzumab govitecan; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sacituzumab Govitecan and Pembrolizumab (Experimental): * Neoadjuvant treatment with pembrolizumab and sacituzumab govitecan is given for a total for 4 cycles. Pembrolizumab is administered first on day 1 every cycle. Sacituzumab govitecan is administered second on day 1 and 8 every cycle. The next cycle should start a minimum 14 days after the Day 8 dose.
  * Surgery is to be performed within 4-8 weeks after day 1 of last cycle of neoadjuvant pembrolizumab/SG.
  * Postoperative radiotherapy is recommended for patients with R1/R2 resection.
  * Maintenance treatment with pembrolizumab alone is given for a total for 13 cycles. This is to be started within 4-8 weeks after surgery or within 4 weeks after postoperative radiotherapy.
  Interventions: Drug: Sacituzumab Govitecan; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Sacituzumab Govitecan — * 4 cycles, each cycle lasting for 3 weeks
  * 10mg/kg given every day 1 and day 8 each cycle
  * IV infusion
Drug: Pembrolizumab — * 4 cycles, each cycle lasting for 3 weeks in Neoadjuvant phase; after surgery, 13 cycles, each cycle lasting for 3 weeks in Maintenance phase.
  * 200mg fixed dose every day 1 each cycle
  * IV infusion

SUMMARY:
The combination of neoadjuvant immunotherapy plus chemotherapy has recently been shown to improve survival outcome compared to chemotherapy alone and was recently approved for resectable non-small cell lung cancer (NSCLC). Despite so, recurrence risk of NSCLC after surgical resection remains high. Sacituzumab govitecan, a novel antibody drug conjugate, was demonstrated to be clinically active in metastatic NSCLC. This study aims to study the clinical efficacy of sacituzumab govitecan plus immunotherapy in resectable NSCLC. This is a open-label, single arm, multicentre, phase II study. Patients with EGFR/ALK negative, stage II-III (AJCC 8th edition), resectable NSCLC are eligible and will receive 4 cycles of neoadjuvant pembrolizumab plus sacituzumab govitecan, followed by surgical resection of tumour, and then 13 cycles of maintenance pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients, 18 years of age or older, able to understand and give written informed consent
2. Pathologically proven NSCLC
3. Tumour tested negative for EGFR and ALK
4. Measurable disease by CT as per RECIST Version 1.1 criteria by investigator
5. Tumour tissue is available for translational research (preferably histology, cytology allowed)
6. AJCC 8th edition Stage II-III based on the following diagnostic workup and tumour is considered potentially resectable

   * Distant metastasis staging by PET/CT whole body or CT thorax and upper abdomen with contrast
   * Patients with stage IIIB (N2) that is considered potentially resectable by cardiothoracic surgeon may be enrolled
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
8. Adequate haematological values without transfusional or growth factor support within 2 weeks of study drug initiation: haemoglobin ≥ 9.0g/dL, absolute neutrophil count ≥ 1.5 x 10^9/L, platelet count ≥ 100 x 10^9/L
9. Adequate hepatic function: bilirubin ≤ 1.5 x ULN, AST/ALT ≤ 2.5 x ULN
10. Adequate renal function: calculated creatinine clearance ≥ 30 ml/min, according to the formula of Cockcroft-Gault equation
11. Male patients and female patients of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception as described in Appendix V.
12. Patients with HBV (HBsAg +ve) must be on antiviral therapy and have a well-controlled HBV infection as determined by investigator. Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease. Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
13. Patients with known HCV infection (positive hepatitis C antibody) (testing is not mandatory for trial enrolment) must have been treated with antiviral therapy and have undetectable HCV viral load.
14. Willing and able to comply with the requirements and restrictions in this protocol.

Exclusion Criteria:

1. Presence of any distant metastasis
2. Previous or concomitant malignancy within 5 years prior registration with the exception of adequately treated localized non-melanoma skin cancer or cervical carcinoma in situ. Prior anti-cancer treatment can be accepted except for drugs listed in exclusion criteria (3) to (8)
3. Received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to study treatment Day 1
4. Mixed SCLC and NSCLC histology
5. Any previous treatment with a PD-1 or PD-L1 or CTLA4 inhibitor, or another agent directed to stimulatory or coinhibitory T-cell receptor (OX40, CD137, etc)
6. Any previous treatment with sacituzumab govitecan, topoisomerase inhibitor, or TROP-2 targeted therapy.
7. Previous radiotherapy to the chest including radiation to mediastinal tumours (e.g. germ cell tumours and thymic tumours)
8. Positive pregnancy test by urine or serum (Appendix V) or women who are breastfeeding
9. Known hypersensitivity to pembrolizumab or Sacituzumab govitecan, or their metabolites or formulation excipient
10. Requirement for ongoing therapy with or prior use of any prohibited medications listed in Appendix IV
11. Absolute contraindications for the use of corticosteroids as premedication
12. Concurrent treatment with other experimental drugs or other anticancer therapy, treatment in a clinical trial within 30 days prior to registration
13. Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment
14. Current or prior use of immunosuppressive medication within 28 days before the first dose of pembrolizumab or sacituzumab govitecan, with the exceptions of intranasal and inhaled corticosteroid or systemic corticosteroids at physiological doses (i.e. which must not exceed 10mg/day of prednisone or an equivalent corticosteroid) and the premedication for chemotherapy.
15. Severe or uncontrolled cardiac disease, congestive heart failure NYHA class III or IV, unstable angina pectoris, history of myocardial infarction during the last 3 months, serious arrhythmias requiring medication (with the exception of atrial fibrillation or paroxysmal supraventricular tachycardia under medical control); history of QTc interval prolongation
16. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illness including, but not limited to, any underlying pulmonary disorder (ie pulmonary embolism within 3 months of enrolment, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc.); history of (non-infectious) pneumonitis that required steroids or recurrent pneumonitis; any autoimmune/connective tissue/inflammatory disorders with pulmonary involvement, or prior pneumonectomy.
17. Active autoimmune disease requiring systemic treatment within the past 2 years or a documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents with the exception of resolved childhood asthma/atopy, hypothyroidism or adrenal insufficiency on hormone replacement, diabetes mellitus stable on insulin replacement
18. Active HBV or HCV infection
19. Known history of Human Immunodeficiency Virus (HIV).
20. History of primary immunodeficiency
21. History of allogeneic organ transplant
22. Receipt of live attenuated vaccination any time during trial therapy and within 30 days of receiving the last dose of trial therapy. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed. COVID-vaccination is allowed.
23. Any concomitant drugs contraindicated for use with pembrolizumab or sacituzumab govitecan including systemic corticosteroid, methotrexate, azathioprine, TNF-alpha blockers.
24. Any other serious underlying medical, psychiatric, psychological, familial condition that in the judgement of the investigator, that may interfere with planned staging, treatment and follow up, affect patient compliance, or place the patient at high risk from treatment-related complications.
25. Patients who refuse surgical treatment of the lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate in the intention-to-treat population | 2 years

SECONDARY OUTCOMES:
Resection rate after neoadjuvant SG and pembrolizumab combination: proportion of patients who undergo surgery with curative intent | 2 years
pCR rates in patients who undergo surgery | 2 years
Major pathological response (MPR) rate in the ITT population and in patients who undergo surgery: MPR is defined as less than 10% viable tumor cells in resected primary tumour specimen | 2 years
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 while on neoadjuvant SG and pembrolizumab combination | 2 years
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 while on adjuvant pembrolizumab | 2 years
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 first 30 days after surgery | 2 years
Objective response rate (ORR): rate of partial and complete response on CT scans according to RECIST criteria ver 1.1 | 2 years
Overall Survival | 2 years
12 month and 24 month event-free survival (EFS) rate | 2 years
Patient reported quality of life (QOL), as measured by EQ-5D-3L during study treatment. | 2 years
  For the descriptive system of EQ-5D-3L, three levels of problems are described in each dimension. For the Visual Analogue Scale (VAS), the overall health assessment of the respondent is captured, ranging from 0 (worst health imaginable) to 100 (best health imaginable)

CONTACTS AND LOCATIONS:
Locations (4):
- Hong Kong (4):
  - Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong
  - Department of Clinical Oncology, Queen Elizabeth Hospital, Hong Kong
  - Department of Clinical Oncology, Tuen Mun Hospital, Hong Kong
  - Department of Oncology, Princess Margaret Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No